CLINICAL TRIAL: NCT07057609
Title: Bioequivalence and Safety Study of Propofol Medium and Long Chain Fat Emulsion Injection in Healthy Chinese Subjects : A Randomized, Open-label, Single-dose, Cross-over Study
Brief Title: Bioequivalence Study of Propofol Medium and Long Chain Fat Emulsion Injection in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HSK-54-BE-2018
Record Dates: First submitted 2025-06-30; First posted 2025-07-10 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test formulation (Experimental): Propofol Medium and Long Chain Fat Emulsion Injection (20 mL:0.2g) Manufacturer: Haisco Pharmaceutical Group Co., Ltd
  Interventions: Drug: Tested Propofol Medium and Long Chain Fat Emulsion Injection (T)
- Reference formulation (Experimental): Propofol Medium and Long Chain Fat Emulsion Injection (20 mL:0.2g) Manufacturer: Fresenius Kabi Deutschland GmbH
  Interventions: Drug: Reference Propofol Medium and Long Chain Fat Emulsion Injection (R)

INTERVENTIONS:
Drug: Tested Propofol Medium and Long Chain Fat Emulsion Injection (T) — Single-dose intravenous infusion of the test formulation under fasting conditions at 30 μg/kg/min. Infusion time: 30 minutes. Dosage: 900 μg/kg for both administrations
  Arms: Test formulation
Drug: Reference Propofol Medium and Long Chain Fat Emulsion Injection (R) — Single-dose intravenous infusion of the reference formulation under fasting conditions at 30 μg/kg/min. Infusion time: 30 minutes. Dosage: 900 μg/kg for both administrations
  Arms: Reference formulation

SUMMARY:
This study assessed the bioequivalence and safety of a single dose of Propofol Medium/Long Chain Fat Emulsion Injection (Test product, Haisco Pharmaceutical Group Co., Ltd.) compared to the reference product (Propofol Medium/Long Chain Fat Emulsion Injection, Fresenius Kabi Deutschland GmbH) in healthy Chinese subjects. Additionally, the pharmacodynamic profiles of both formulations were evaluated

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Chinese male or female participants aged 18-55 years (inclusive).
2. Body weight ≥50.0 kg (male) or ≥45.0 kg (female), with a body mass index (BMI) of 19.0-26.0 kg/m² (inclusive).
3. No potential difficult airway or loose teeth.
4. No history of anesthesia-related complications or adverse events.
5. Normal or clinically nonsignificant findings in: physical examination, vital signs, laboratory tests (including complete blood count, urinalysis, blood biochemistry, coagulation profile, and pregnancy test for all females), 12-lead electrocardiogram (ECG), eligibility confirmed by the investigator despite minor abnormalities.
6. Participants (and their partners) agree to use effective contraception and avoid pregnancy plans from signing the informed consent form until 3 months after the last dose of the investigational product.
7. Capable of comprehending study procedures, willing to provide written informed consent, and able to comply with the trial protocol.

Exclusion Criteria:

1. History or presence of clinically significant diseases affecting major systems (e.g., digestive, respiratory, urinary, cardiovascular, endocrine, neurological, hematological, immunological, psychiatric, or metabolic disorders), familial genetic disorders, or any condition deemed by the investigator to interfere with study outcomes.
2. Severe infection, trauma, or major surgery within 4 weeks prior to screening, or planned surgical procedures during the study period.
3. History of drug abuse (e.g., chronic use of NSAIDs, opioids, sedatives, or addictive substances) within 12 months prior to screening, or positive urine drug screen.
4. Hypersensitivity (e.g., drug/food allergies) or known allergy to propofol or excipients in propofol medium/long-chain triglyceride emulsion (e.g., soybean oil, medium-chain triglycerides, egg lecithin, glycerol, oleic acid, sodium hydroxide).
5. Excessive alcohol consumption (defined as >14 units/week; 1 unit = 360 mL beer, 45 mL 40% spirits, or 150 mL wine) within 6 months prior to screening, positive alcohol test, or unwillingness to abstain from alcohol during the study.
6. Smoking >5 cigarettes/day within 3 months prior to screening or inability to abstain from smoking during the study.
7. Use of prescription drugs, over-the-counter (OTC) medications, supplements (including vitamins), or herbal remedies within 2 weeks prior to screening.
8. Participation in another clinical trial within 3 months prior to screening, ongoing follow-up in another study, or planned enrollment in other trials during this study.
9. History or current diagnosis of autonomic dysfunction (e.g., recurrent syncope, palpitations) within the past 3 years.
10. Severe sleep apnea syndrome.
11. Positive serological tests for HBsAg, HCV antibodies, Treponema pallidum antibodies, or HIV antibodies.
12. Family history of malignant hyperthermia.
13. Hemophobia, needle phobia, or inability to tolerate venipuncture.
14. Lactating females or positive pregnancy test during screening or the study period.
15. Dietary restrictions incompatible with study center meals or protocol requirements.
16. Consumption of specific foods/beverages (e.g., grapefruit, xanthine-containing products) or substances affecting drug ADME (absorption, distribution, metabolism, excretion) within 48 hours prior to dosing.
17. Any other condition deemed by the investigator to compromise subject safety or data validity.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2019-03-22 (Actual)

PRIMARY OUTCOMES:
Cmax | From the start of intravenous infusion to 480 minutes after the intravenous infusion
  The maximum blood concentration, the pharmacokinetic parameters of Propofol in plasma
AUC(0-t) | From the start of intravenous infusion to 480 minutes after the intravenous infusion
  The area under the blood concentration-time curve from time 0 to the last accurately measurable concentration at sample collection time t was measured, the pharmacokinetic parameters of Propofol in plasma
AUC(0-∞) | From the start of intravenous infusion to 480 minutes after the intravenous infusion
  The area under the blood concentration-time curve from 0 to infinite time (∞), the pharmacokinetic parameters of Propofol in plasma

SECONDARY OUTCOMES:
BIS AUC0-60min | From the start of intravenous infusion to 60 minutes after the intravenous infusion
  Area under the BIS positive peak-time curve from 0 to 60 minutes after converting the BIS value to a positive peak (100-BIS)
BISmin | From the start of intravenous infusion to 60 minutes after the intravenous infusion
  Minimum BIS value
t-BISmin | From the start of intravenous infusion to 60 minutes after the intravenous infusion
  Time to reach the minimum BIS value
AEs | From the time of signing ICF to the end of follow-up，up to 10 days
  The incidence and severity of AEs

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China